CLINICAL TRIAL: NCT05904119
Title: Lomustine With and Without Reirradiation for First Progression of Glioblastoma: a Randomized Phase III Study
Acronym: LEGATO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2227-BTG
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: First Progression of Glioblastoma
Keywords: First progression; Glioblastoma; Phase III; Lomustine; Reirradiation
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Lomustine alone
  Interventions: Drug: Lomustine
- Experimental group (Experimental): Lomustine plus reirradiation
  Interventions: Drug: Lomustine; Radiation: Reirradiation

INTERVENTIONS:
Drug: Lomustine — Oral administration of Lomustine
Radiation: Reirradiation — Given at least 6 months after the end of prior radiotherapy
  Arms: Experimental group

SUMMARY:
Despite comprehensive multimodal treatment of newly diagnosed glioblastoma, almost all patients suffer from tumour relapse. Currently, no standard of care exists to treat these tumour relapses. Treatment options include repeated surgery (if feasible), systemic therapy (bevacizumab, lomustine, temozolomide re-challenge), reirradiation and best supportive care. Currently, the superiority of combined chemoradiation versus chemotherapy alone remains unproven. Given that lomustine is the standard chemotherapeutic agent for the treatment of recurrent glioblastoma in Europe and the unclear efficacy of reirradiation, we want to explore whether combining lomustine and reirradiation may be a better treatment than lomustine alone. The results of the prospective randomized trial proposed here should demonstrate a significant improvement in overall survival when lomustine is combined with reirradiation in patients with recurrent glioblastoma compared to lomustine alone without adversely affecting quality of survival. The trial will be stopped based on overall survival in a preplanned futility and efficacy interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Before patient's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Patients with first progression or recurrent glioblastoma after standard chemoradiotherapy (any treatment other than use of nitroureas) having occurred at least 6 months after the end of prior radiotherapy
* Measurable disease according to RANO criteria with a maximum tumour diameter of 5 cm (local investigator assessment)
* In case of surgery for recurrence: fully recovered from surgery, confirmation of recurrence by histology, and patient fit for treatment as per local investigator assessment.
* Histologically proven diagnosis of glioblastoma, IDH wildtype per WHO 2021 classification and local assessment of tissue from diagnosis or recurrence
* Initial treatment of newly diagnosed glioblastoma by maximal safe resection and postsurgical concurrent conventionally fractionated or abbreviated (minimum 15 fractions) chemoradiotherapy with or without maintenance chemotherapy with temozolomide (patient must have received at least one dose)
* Stable or decreasing dose of steroids for 7 days prior to enrolment
* Age ≥ 18 years
* WHO Performance status of 0-2
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential must agree to use adequate birth control measures during the study treatment period and for at least 6 months after the last dose of study treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Non-sterile males must use contraception during treatment and for 6 months after the last dose.
* Non-sterile males must avoid sperm donation for the duration of the study and for at least 6 months after the last dose of study treatment.

Exclusion Criteria:

* Any prior anticancer treatment for recurrent glioblastoma (except surgery)
* Significant reduction in thrombocyte and/or leukocyte counts as well as severe renal impairment according to investigator's opinion
* History or present acute leukaemia or any myeloid disease
* Known hypersensitivity to the active components or excipients of lomustine
* Known coeliac disease or wheat allergy
* Live attenuated vaccine in the 3 months prior to lomustine initiation
* Any serious or uncontrolled medical condition (e.g., infections, chronic alcoholism, drug addiction) or abnormality, in the judgment of the investigator that prohibits obtaining informed consent, safe participation and study completion
* Known contraindication to imaging tracer or any product of contrast media and Magnetic Resonance Imaging (MRI) contraindications
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of enrolment up to the date of death, assessed up to 40 months after first patient is enrolled
  Defined as the number of days from date of enrolment to the date of death due to any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the date of enrolment up to the date of first objective progression or the date of death whichever occur first, assessed up to 40 months after first patient is enrolled
  Events are progressions based on Response Assessment in Neuro Oncology (RANO) criteria as determined by the local investigator .
Health-related Quality of Life (HRQoL) | From the date of enrolment until disease progression, assessed up to 40 months after first patient is enrolled
  HRQoL will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3.
Toxicity profile of lomustine plus reirradiation | From the date of enrolment until end of study treatment 30 (± 7 days) after last dose, assessed up to 40 months after first patient is enrolled
  Safety according to the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for toxicity and Serious Adverse Event reporting.
Neurocognitive functioning of lomustine pus reirradiation | From the date of enrolment until end of study treatment 30 (± 7 days) after last dose, assessed up to 40 months after first patient is enrolled
  Neurocognitive functioning assessed by Mini Mental State Examination (MMSE)
To transform self-reported quality of life data from the QLQ-C30 into health utility values, ready to be used in subsequent health economic analyses. | From the date of enrolment until disease progression, assessed up to 40 months after first patient is enrolled
  A deterioration event is defined as ≥>10-point worsening from baseline in the GHQ without further improvement (i.e., no subsequent ≥>10 point improvement) or death due to any cause.
Objective response (ORR) | From the date of enrolment up to the date of first objective progression or the date of death whichever occur first, assessed up to 40 months after first patient is enrolled
Complete response (CRR) | From the date of enrolment up to the date of first objective progression or the date of death whichever occur first, assessed up to 40 months after first patient is enrolled

OTHER OUTCOMES:
To assess health-related quality of life over time based on the results of 3 different scales (QLQ-C30, QLQ-BN20 and the item list (IL46)). | From the date of enrolment until disease progression, assessed up to 40 months after first patient is enrolled
  Changes in HRQoL from baseline in the GHQ/QoL, fatigue, nausea/vomiting, physical, role and social functioning scale scores assessed over time will be evaluated descriptively. Descriptive summaries such as median, range (minimum, maximum), IQR, mean and standard deviation will be provided for all the other scales from the QLQ-C30, QLQ-BN20 and the item list (IL46).
  For functional and global HRQoL scales, higher scores represent a better level of functioning and are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represents more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, Prof., Principal Investigator — EORTC Study Coordinator; Giuseppe Minniti, Dr., Principal Investigator — EORTC Study Coordinator
Locations (42):
- Austria (3):
  - A.O Landeskrankenhaus - Innsbruck Universitaetsklinik, Innsbruck
  - Kepler University Hospital - Neuromed campus, Linz
  - Universitaetsklinikum Wien - AKH unikliniken, Vienna
- Belgium (4):
  - AZORG, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi - Site Les Viviers, Gilly
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Masaryk Memorial Cancer Institute, Brno, Czechia
- Aarhus University Hospitals - Region Midtjylland - Aarhus University Hospital-Skejby, Aarhus, Denmark
- France (9):
  - CHU d'Amiens - CHU Amiens Picardie - Site Sud, Amiens
  - CLCC - Jean Perrin, Clermont-Ferrand
  - CHRU de Lille, Lille
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - CHU de Nice - Hôpital Pasteur, Nice
  - Assistance Publique Hopitaux Paris- APHP - APHP Sorbonne Univ - Hopital la Pitie-Salpetriere (233), Paris
  - Assistance Publique Hopitaux Paris- APHP - APHP Nord - Univ De Paris Cite - Hop. Saint Louis, Paris
  - Institut de Cancerologie de l´Ouest (ICO) - Saint Herblain, Saint-Herblain
- Germany (8):
  - Univ. Knappschaft Krankenhaus Bochum, Bochum
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Erlangen-Schwabachanlage, Erlangen
  - Universitaetsklinikum Heidelberg - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitätsklinikum Leipzig-Klinik für Strahlentherapie und Radioonkologie, Leipzig
  - Ludwig-Maximilians-Universitaet Muenchen - Campus Grosshadern, Munich
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen- Crona Kliniken, Tübingen
- Italy (5):
  - IRCCS-Ospedale Bellaria-Bologna, Bologna
  - ULSS 9 Scaligera Veneto - Azienda Unita Locale Socio-Sanitaria N. 9-Mater Salutis Hospital, Legnago
  - Istituto Clinico Humanitas, Milan
  - IRCCS - Istituto Oncologico Veneto, Padua
  - Azienda ospedaliero Univ Policlinico Umberto I, Roma
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, Rotterdam
  - ETZ Tilburg - ETZ - St. Elisabethziekenhuis, Tilburg
- Norway (2):
  - Oslo University Hospital - Radiumhospitalet, Oslo
  - St Olavs University Hospital - St. Olavs Hospital, Trondheim University Hospital, Trondheim
- Spain (4):
  - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia) (381), Badalona
  - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
- Oncology Institute of Southern Switzerland (IOSI) - Ospedale San Giovanni, Bellinzona, Switzerland

REFERENCES:
- [Derived] Preusser M, Kazda T, Le Rhun E, Sahm F, Smits M, Gempt J, Koekkoek JA, Monti AF, Csanadi M, Pitter JG, Bulbek H, Fournier B, Quoilin C, Gorlia T, Weller M, Minniti G; European Organisation for Research, Treatment of Cancer (EORTC) Brain Tumor Group. Lomustine with or without reirradiation for first progression of glioblastoma, LEGATO, EORTC-2227-BTG: study protocol for a randomized phase III study. Trials. 2024 Jun 7;25(1):366. doi: 10.1186/s13063-024-08213-7. PMID 38849943